CLINICAL TRIAL: NCT05663294
Title: Partial Radiotherapy for Breast in Situ Carcinoma of Intermediate Low Risk As Local Adjuvant Treatment
Brief Title: PBI for Breast in Situ Carcinoma of Intermediate Low Risk As Local Adjuvant Treatment
Acronym: PRISCILLA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Mediolanum Cardio Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3271
Record Dates: First submitted 2022-12-05; First posted 2022-12-23 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Partial Breast Irradiation (Experimental): Radiation treatment will be started within 120 days after surgery. The fractionation schedule depends on the policy of the treating center, but is mandatory to use CT-based planning. Both once-daily and twice-daily schedule are allowed.
  The allowed schedules for external beams radiotherapy are:
  * 40 Gy in 15 fractions;
  * 30 Gy in 5 fractions;
  * 40 Gy or 38.5 in 10 twice-daily fractions (each daily dose must be separated by at least 6 hours).
  The schedule for brachytherapy are:
  * 32 Gy in 8 twice-daily fractions for HDR;
  * 30.3 Gy in 7 twice-daily fractions for HDR;
  * 50Gy 0.60-0.80 Gy/hour (1 pulse/hour, 24 hours/day) for PDR.
  Interventions: Radiation: external beams radiotherapy; Radiation: brachytherapy

INTERVENTIONS:
Radiation: external beams radiotherapy — External beam radiation therapy uses high doses of radiation to destroy cancer cells and shrink tumors. A large machine aims radiation at the cancer. The allowed schedules for external beams radiotherapy are:
  * 40 Gy in 15 fractions;
  * 30 Gy in 5 fractions;
  * 40 Gy or 38.5 in 10 twice-daily fractions (each daily dose must be separated by at least 6 hours).
Radiation: brachytherapy — Brachytherapy is a form of radiation therapy where a sealed radiation source is placed inside or next to the area requiring treatment.
  The schedule for brachytherapy are:
  * 32 Gy in 8 twice-daily fractions for HDR;
  * 30.3 Gy in 7 twice-daily fractions for HDR;
  * 50Gy 0.60-0.80 Gy/hour (1 pulse/hour, 24 hours/day) for PDR.

SUMMARY:
Screening and advances in breast imaging led to a continuous increase of Ductal Carcinoma in situ (DCIS) diagnosis. Whole breast radiotherapy was reported to be effective in reducing the risk of local recurrence in all analyzed patients and tumor characteristics. In order to de-escalate treatment in low and intermediate DCIS, it is possible to investigate the role of partial breast irradiation (PBI). To date, data from available literature supports the hypothesis that PBI is a safe well tolerated therapy that appears to be equivalent to WBI in terms of efficacy and ultimate breast cosmesis.

DETAILED DESCRIPTION:
Screening and advances in breast imaging led to a continuous increase of Ductal Carcinoma in situ (DCIS) diagnosis. Unfortunately, the management of this specific disease is still debated regarding adjuvant therapy (radiation therapy and endocrine therapy) after breast conserving surgery (BCS).

Four randomized trials have shown a decrease of the local recurrence (LR) using adjuvant radiotherapy with conventional fractionation (50 Gy in 25 fractions). In the early breast cancer trialists' collaborative Group (EBCTCG) overview (7) radiotherapy approximatively halved the ipsilateral breast event (IBE) rate, from 28.1% to 12.9 % at 10 years. Radiotherapy was reported to be effective in reducing the risk of local recurrence in all analyzed patients and tumor characteristics (e.g. age, tumor size, histological grade, comedonecrosis, etc.), but no differences were seen in distant metastases, breast cancer-specific survival, or overall survival between irradiated and un-irradiated patients. Nowadays, progress in diagnosis and a greater attention in achieving negative surgical margins increased the interest in identifying sub groups of patient in which a treatment de-escalation could be possible. Some prospective randomized and non-randomized trials try to define a low-risk cohort in which radiotherapy could be omitted. RTOG 9804 randomized 711 low-intermediate risk patients to RT versus nothing and find that LF rate decreased significantly with the addition of RT.

De-escalation of radiation therapy treatment could be done with partial breast irradiation (PBI). In modern era 7 randomized trials analyzed the efficacy of PBI versus whole breast RT in low-risk patients with early stage breast cancer, using different techniques. Those studies drive ESTRO and ASTRO to endorse the use of PBI out of clinical trials. In general, PBI involves treating the surgical cavity with a 1- to 2-cm margin, thus reducing the volume of treated breast tissue by up to 50% using various methods. Technical approaches of PBI include multicatheter interstitial brachytherapy, balloon catheter brachytherapy, external 3-D conformal external beam radiotherapy (3D-CRT), intensity modulated radiotherapy (IMRT) and intraoperative radiotherapy (IORT). Park et al. reported a retrospective study on 53 patients treated with MammoSite brachytherapy or 3D-CRT, with a Three-year actuarial ipsilateral breast tumor recurrence was 2%. Becherini et al. analyzed the long-term efficacy and safety results of the series of 22 patients with DCIS enrolled in the accelerated PBI arm of the APBI-IMRT-Florence phase 3 trial and found 5- and 10-year local recurrence, distant metastasis-free survival, and breast cancer-specific survival of 100%.

To date, data from available literature supports the hypothesis that PBI is a safe well tolerated therapy that appears to be equivalent to WBI in terms of efficacy and ultimate breast cosmesis in infiltrating carcinoma. Data on DCIS are missing.

Based on this background, we designed a study to evaluate 5-year Local Control rate of Partial Breast Irradiated (PBI) using external beam radiotherapy (3D-CRT, VMAT-RA, Tomotherapy or Cyberknife) or brachytherapy in a selected group of women with low-intermediate DCIS.

ELIGIBILITY:
Inclusion Criteria:

* Age >40
* Pathologically confirmed DCIS:

  1. low risk (lesions of ≤3 cm diameter, resection margins of at least 2 mm, nuclei grade: G1, G2)
  2. intermediate risk (lesions of ≤1 cm diameter, resection margins of at least 2 mm, nuclei grade: 3)
* Written informed consent

Exclusion Criteria:

* Prior thoracic radiation therapy
* Preoperative systemic treatments (i. e., chemotherapy, endocrine therapy);
* Autoimmune disease, vasculitis, collagenopathy or scleroderma that may predispose to late sequelae
* No other cancers in the last 5 years

Min Age: 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Local Control rate | 5 years
  Absence of the occurrence of new lump in the irradiated breast or appearance of skin lesions; it will be divided in inside or outside the treated area, evaluating the localization in the breast. For the evaluation it will be used bilateral mammography.

SECONDARY OUTCOMES:
toxicities assessed by "Common Terminology Criteria for Adverse Events (CTCAE) v5.0" | 5 years
  Evaluation of toxicities due to partial breast irradiation, toxicities grade and specific term will be given using "Common Terminology Criteria for Adverse Events (CTCAE) v5.0".
The Harvard Scale | 5 years
  aesthetic evaluation after partial breast irradiation. Cosmesis will be evaluated using The Harvard Scale of cosmetic outcome. The results will be % of the 4 possible outcomes (Excellent, Good, Fair, Poor)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Clinico Humanitas, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided